CLINICAL TRIAL: NCT05145985
Title: Senior Fitness Test - Proposed Reference Curves for Polish Women Over 60
Brief Title: Senior Fitness Test - Reference Curves for Polish Women Over 60
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: SFT-2021
Record Dates: First submitted 2021-10-14; First posted 2021-12-06 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Aging; Physical Fitness
Keywords: aged; physical fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women over 60: Women aged over 60 years. Participants were allowed to participate in the study if they were able to walk independently and their health condition allowed them to perform the indicated fitness tests.
  Interventions: Diagnostic Test: Senior Fitness Test

INTERVENTIONS:
Diagnostic Test: Senior Fitness Test — Senior Fitness Test is comprised of 6 individual test items and for a description of the trials. All fitness tests (1-6) were selected for analysis:
  1. Arm Curl (AC) - measurement of upper body muscle endurance - numbers of arm curls as possible in 30 seconds (n)
  2. 30-second Chair Stand (30SCS) - measurement of lower body strength; numbers of chair stand as possible in 30 seconds (n)
  3. Back Scratch Test (BST) - measurement of upper-body flexibility; the best score to the nearest centimeter (cm)
  4. Chair Sit and Reach Test (CSRT)- measurement of lower-body flexibility (specifically hamstring flexibility); the best score to the nearest centimeter (cm)
  5. 8-Foot Up and Go (TUG) - measurement of agility (dynamic balance) and aerobic endurance; the best time of the two trails to the nearest 1/10th second (s)
  6. 2-Minute Walk Test (2MWT) - measurement of (aerobic) endurance; the total number of times the right knee reaches the tape level in two minutes (n)

SUMMARY:
The aging of society is a natural process, but it entails challenges in social, economic and health aspects. It is important for mature people to maintain, for as long as possible, adequate functional capacity to live independently and autonomously. Presentation of reference values of functional abilities in continuous perspective (and not in 5-year periods as it is in standards for SFT) is a better approach. This approach reflects the process of change that occurs in functional ability. The aim of the study was to develop centile distributions of fitness tests constituting the Senior Fitness Test (SFT) for women over 60 years of age in Poland, moving independently.

DETAILED DESCRIPTION:
The aging of society is a natural process, but it entails challenges in social, economic and health aspects. It is important for mature people to maintain, for as long as possible, an adequate functional capacity to live independently and autonomously. In order to determine the level of functional fitness, fitness tests are used. Such tests include the Senior Fitness Test (another name: Fullerton Functional Fitness Test)- tests described below; One Leg Standing Test - test that assesses static balance to diagnose symptoms of mobility disability; Stops Walking When Talking - assesses risk of falling and ability to perform two activities simultaneously (talking and walking), Berg Balance Scale - assesses ability to maintain balance while performing specific tasks, does not assess gait; Four Square Step Test (FSST) - assesses dynamic balance and coordination; Functional Reach Test (FRT) - oceans of dynamic balance; Tinetti Test - oceans of balance during simple tasks and oceans of gait; Short Physical Performance Battery - oceans of balance functioning and lower limb performance in people over 60. age. On the basis of these fitness tests the level of a selected aspect of functional ability is assessed, converting the results into points. Among the indicated tools the Senior Fitness Test seems to be the most universal, as it is a comprehensive and useful tool for multidimensional assessment of physical fitness of people over 60. It allows observation of the gradual decline in functional ability with age. Additionally, the simple tests and norms for the fitness tests in the Senior Fitness Test are defined for people aged 60-94. Publicly available norms were developed for the American population.

The development of reference values for the fitness tests that make up the Senior Fitness Test reflects the process that is taking place in the functional fitness area of people over 60 years of age. Additionally it is possible to observe changes on a continuous basis rather than in 5-year periods. It also allows to catch the moment when functional fitness deterioration occurs.

The main objective was to develop centile grids for fitness tests assessing upper and lower limb muscle strength, flexibility, dynamic balance and endurance, which comprise the Senior Fitness Test for women over 60.

The Senior Fitness Test is a tool used to determine the functional fitness level of people over 60 years of age. In order to determine physical fitness levels, Senior Fitness Test was carried out. The test is comprised of 6 individual test items and for a description of the trials, please refer to Różańska-Kirschke et al. All fitness tests (1-6) were selected for analysis:

1. Arm Curl (AC) - measurement of upper body muscle endurance.
2. 30-second Chair Stand (30SCS) - measurement of lower body strength.
3. Back Scratch Test (BST) - measurement of upper-body flexibility.
4. Chair Sit and Reach Test (CSRT) - measurement of lower-body flexibility (specifically hamstring flexibility)
5. 8-Foot Up and Go (TUG) - measurement of agility (dynamic balance) and aerobic endurance.
6. 2-Minute Walk Test (2MWT) - measurement of (aerobic) endurance.

ELIGIBILITY:
Inclusion Criteria:

* gender - female
* age - over 60
* able to move independently
* health condition allowing to perform the agility tests
* consent to participate in the study

Exclusion Criteria:

* age - under 60
* unable to move around independently
* health condition does not allow you to take part in the fitness tests
* no consent to participate in the study

Ages: 60 Years to 94 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consisted of all individuals who will to participate in the study and meet the specified inclusion conditions.
Sampling Method: Non-Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
determining the level of fitness in individual fitness tests - measure leg strength | baseline
  1. The chair stand test - number of completed chair stands in 30 seconds (n) This test assesses leg strength and endurance. Equipment: a straight back or folding chair without arm rests (seat 44 cm high) Test: Place the chair against a wall, or otherwise stabilize it for safety. The subject sits in the middle of the seat, with their feet shoulder width apart, flat on the floor. The arms are to be crossed at the wrists and held close to the chest. From the sitting position, the subject stands completely up, then completely back down, and this is repeated for 30 seconds. Count the total number of complete chair stands (up and down equals one stand). If the subject has completed a full stand from the sitting position when the time is elapsed, the final stand is counted in the total (from Jones & Rikli, 2002).
determining the level of fitness in individual fitness tests - measure upper body strength | baseline
  2. The Arm Curl test - the total number of controlled arm curls performed in 30 seconds (n) Equipment: 2kg weight, a chair without armrests, stopwatch. Test: do as many arm curls as possible in 30 seconds. This test is conducted on the dominant arm side (or stronger side). The subject sits on the chair, holding the weight in the hand using a suitcase grip (palm facing towards the body) with the arm in a vertically down position beside the chair. Brace the upper arm against the body so that only the lower arm is moving (tester may assist to hold the upper arm steady). Curl the arm up through a full range of motion, gradually turning the palm up (flexion with supination). As the arm is lowered through the full range of motion, gradually return to the starting position. Repeat this action as many times as possible within 30 seconds.
determining the level of fitness in individual fitness tests - measure lower body flexibility | baseline
  3. The Chair Sit and Reach test - The score is recorded to the nearest 0,5 cm or 1 cm as the distance reached, either a negative or positive score (cm) Equipment: ruler, straight back or folding chair (about 44 cm high) Test: The subject sits on the edge a chair (placed against a wall for safety). One foot must remain flat on the floor. The other leg is extended forward with the knee straight, heel on the floor, and ankle bent at 90°. Place one hand on top of the other with tips of the middle fingers even. Instruct the subject to inhale, and then as they exhale, reach forward toward the toes by bending at the hip. Keep the back straight and head up. The distance is measured between the tip of the fingertips and the toes. Measure the distance between the fingers and the toes (a negative score), if they overlap, measure by how much (a positive score).
determining the level of fitness in individual fitness tests - measure general shoulder range of motion | baseline
  4. The Back Scratch Test - Record the best score to the nearest centimeter or 0,5 cm. The higher the score the better the result (cm) This test is done in the standing position. Place one hand behind the head and back over the shoulder, and reach as far as possible down the middle of your back, your palm touching your body and the fingers directed downwards. Place the other arm behind your back, palm facing outward and fingers upward and reach up as far as possible attempting to touch or overlap the middle fingers of both hands. An assistant is required to direct the subject so that the fingers are aligned, and to measure the distance between the tips of the middle fingers. If the fingertips touch then the score is zero. If they do not touch, measure the distance between the finger tips (a negative score), if they overlap, measure by how much (a positive score).
determining the level of fitness in individual fitness tests - measure speed, agility and balance while moving | baseline
  5. The '8 Foot Up-and-Go' test - Take the best time of the two trails to the nearest 1/10th second (s) equipment: stopwatch, straight back or folding chair (44 cm high) Test: Place the chair next to a wall (for safety) and the marker 8 feet in front of the chair. Clear the path between the chair and the marker. The subject starts fully seated, hands resting on the knees and feet flat on the ground. On the command, "Go," timing is started and the subject stands and walks (no running) as quickly as possible (and safely) to and around the cone, returning to the chair to sit down. Timing stops as they sit down.
determining the level of fitness in individual fitness tests - measure aerobic endurance | baseline
  6. The 2-Minute Step in Place test - Record the total number of times the right knee reaches the tape level in two minutes (n) equipment: tape for marking the wall, stopwatch Test: The subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the patella (knee cap) and illiac crest (top of the hip bone). The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed, and holding onto the wall or a stable chair is allowed. Stop after two minutes of stepping.

CONTACTS AND LOCATIONS:
Locations (1):
- the Józef Piłsudski University of Physical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided